CLINICAL TRIAL: NCT01795105
Title: Post-Marketing Surveillance of Safety and Efficacy of Abilify® Tablets in Korean Patients With Tourette's Disorder Under the "New Drug Re-Examination"
Brief Title: ABF Tourette's Disorder Post Marketing Surveillance Study
Status: Completed | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 031-KOA-1101n
Record Dates: First submitted 2013-01-31; First posted 2013-02-20 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-01

CONDITIONS: Tourette's Disorder
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Aripiprazole (Abilify® Tablets/Abilify® ODT)

SUMMARY:
This is a Post-Marketing Surveillance study of Abilify® tablets in accordance with Korean regulations on New Drug Re-examination (i.e. New Drug Re-examination Standards: KFDA Notification No. 2010-94 dated 27 December 2010).

DETAILED DESCRIPTION:
This study will be conducted in a prospective, single-arm, multi-center format. As this study is observational in nature, the patient's follow-up is not prescriptive in nature and must be left up to the judgment of the physician (investigator), within the period of observation set forth in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 6 to 18 years of age with Tourette's Disorder
* Patients who are prescribed Abilify® treatment as per investigator's medical judgment.
* Patients who gave written authorization to use their personal and health data
* Patients starting Abilify® treatment after agreement is in place

Exclusion Criteria:

* Patients with known hypersensitivity to Aripiprazole or any excipients of Abilify®
* Patients who have been treated with Abilify®
* Patients with rare hereditary problems of galactose intolerance, the lapp lactase deficiency, or glucose-galactose malabsorption
* Patients with score 0(Not assessed) or 1(Normal, not at all ill) in the TS-CGI-S
* Patients participating in other clinical trial

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients 6 to 18 years of age with Tourette's Disorder according to the approved product market authorization
Sampling Method: Probability Sample
Enrollment: 692 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05-29 (Actual); Study Completion 2015-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Seoul
  - Seoul Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole (Abilify® Tablets/Abilify® ODT): 1. Pediatric patients 6 to 18 years of age with Tourette's Disorder
  2. Patients who are prescribed Abilify® Tablets/Abilify® ODT treatment as per investigator's medical judgment.
  3. Dose: Aripiprazole (Abilify® Tablets 2mg, 5mg, 10mg, 15mg, Abilify® ODT 10mg, 15mg)
Period: Overall Study
Arm/Group | Aripiprazole (Abilify® Tablets/Abilify® ODT)
Started | 692
Completed | 648
Not Completed | 44

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole (Abilify® Tablets/Abilify® ODT): Pediatric patients with Tourette syndrome aged 6-18 years who were administered with Aripiprazole (Abilify® Tablets/Abilify® ODT) according to the approved dosage.
Arm/Group | Aripiprazole (Abilify® Tablets/Abilify® ODT)
Number analyzed (Participants) | 648
Age, Customized [Count of Participants; unit: Participants]
  >=6 years and <12 years | 449
  >=12 years and <18 years | 199
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex information of 1patient haven't been examined although we asked inversigater to resolve the query.So, it is missing value.
  Participants
    number analyzed (Participants) | 647
    Female | 114
    Male | 533

OUTCOME MEASURES:

1. Primary Outcome: Frequency (n) of Subjects With Adverse Event
Description: Frequency (n) and Percentage(%) of subjects with Adverse event
Time Frame: Follow-up at least once from baseline to 6 weeks and at least 12weeks
Measure: Count of Participants; unit: Participants
Groups:
- Aripiprazole Main Surveillance: Patients who were given Abilify Tablet or Abilify OD Tablet for at least 6 weeks or longer.
- Aripiprazole Long-term Surveillance: Patients who were given Abilify Tablet or Abilify OD Tablet for at least 12 weeks.
Arm/Group | Aripiprazole Main Surveillance | Aripiprazole Long-term Surveillance
Number analyzed (Participants) | 648 | 233
Participants
  Number of patients reported for AE | 50 | 19
  Number of patients reported for ADR | 42 | 14

2. Secondary Outcome: Mean Change in the TS-CGI(Tourette's Syndrome-Clinical Global Impression-Improvement)
Description: Mean change in the TS-CGI from baseline to next visit(at least 6, 12 weeks interval from baseline) post-treatment
  *TS-CGI scale 0=Not assessed
  1. Normal, not at all ill
  2. Borderline ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Extremely ill
Time Frame: at least 6, 12 weeks interval from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole Main Surveillance | Aripiprazole Long-term Surveillance
Number analyzed (Participants) | 589 | 233
score on a scale
  at the first visit | 4.31 (0.81) | 4.34 (0.86)
  at the last visit | 2.73 (0.83) | 2.66 (0.80)
  Mean change in the TS-CGI | -1.58 (0.95) | -1.69 (0.93)

ADVERSE EVENTS:
Arm/Group | Aripiprazole (Abilify® Tablets/Abilify® ODT)
Serious Adverse Events (participants affected / at risk) | 1/648
Other Adverse Events (participants affected / at risk) | 49/648
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (Abilify® Tablets/Abilify® ODT) (N=648)
Neuritis (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (Abilify® Tablets/Abilify® ODT) (N=648)
Somnolence (Psychiatric disorders) | 16 (16)
Appetite increased (Psychiatric disorders) | 4 (4)
Anorexia (Psychiatric disorders) | 2 (2)
Apathy (Psychiatric disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 2 (2)
Emotional liability (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (10)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Mouth dry (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 4 (5)
Hyperkinesia (Nervous system disorders) | 3 (3)
Hypertonia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weight increase (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2014-02-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT01795105/Prot_000.pdf